CLINICAL TRIAL: NCT02381145
Title: Long-term Supplementation of Dietary Polyphenols as Modulators of Lipid Oxidation and Mitochondrial Function in Overweight Volunteers
Brief Title: Dietary Polyphenols and Insulin Sensitivity in Overweight and Obese Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NL31421.068.10
Record Dates: First submitted 2013-08-20; First posted 2015-03-06 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Healthy
Keywords: Polyphenols; Resveratrol; Epigallocatechin-gallate; Insulin sensitivity; mitochondrial function; lipid oxidation; tissue lipolysis
MeSH Terms: conditions — Insulin Resistance | interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): micro-cellulose-filled Placebo
  Interventions: Dietary Supplement: Placebo
- EGCG+RSV-supplementation (Active Comparator): EGCG+RSV: 300mg/d + 80mg/d
  Interventions: Dietary Supplement: EGCG+RSV-supplementation

INTERVENTIONS:
Dietary Supplement: EGCG+RSV-supplementation — Teavigo (~300mg/d) Resveratrol (~80mg/d)
  Other Names: Teavigo, Pure Encapsulations Inc. (Massachusetts, USA); Resveratrol, Pure Encapsulations Inc. (Massachusetts, USA)
  Arms: EGCG+RSV-supplementation
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
In this double-blind, randomized, placebo-controlled study, we aim to investigate the effects of a long-term supplementation on insulin sensitivity, mitochondrial function and substrate metabolism in healthy overweight men and women.

In each group, 21 subjects consume 100mg Resveratrol (RSV) and 150mg Epigallocatechin-gallate (EGCG), respectively Placebo capsules, twice daily over a period of 12 weeks. The subjects receive the capsules after the last pre-measurement and continue to take them throughout the post-measurements.

Before and after the supplementation period, we perform a hyperinsulinemic-euglycemic clamp with a glucose-tracer infusion to assess hepatic and systemic insulin sensitivity. Simultaneously, substrate oxidation is measured throughout the clamp by indirect calorimetry. Furthermore, we perform a high-fat mixed meal test, in which we collect blood and measure substrate oxidation during fasted and postprandial conditions. During the meal tests, extra plasma is collected at the start (t=-30) and the end (t=240), of which the supernatant is stored in light-protected tubes (EGCG is mixed 1:1 with an EGCG buffer) for analyzing polyphenol concentrations in the blood.

In the male subgroup (21 men), we additionally place each 2 microdialysis probes in the subcutaneous adipose tissue and the gastrocnemius in order to assess local lipolysis and blood flow by means of ethanol infusion.

Furthermore, a dexa-scan is performed to assess body composition and biopsies are taken under fasted conditions from the subcutaneous adipose tissue and the quadriceps femoralis muscle. These samples are stored at -80C. Part of the adipose tissue samples is collected to measure adipocyte size. Of the skeletal muscle biopsy, one part is directly buffered and used for the oxygraph to measure mitochondrial function.

At last, feces samples are collected before and after the intervention in order to assess energy content, microbial composition and short-chain fatty acid content.

Based on previous human studies in our and other departments, we hypothesize that after 12 weeks of the combined polyphenol supplementation, insulin sensitivity and mitochondrial function improve. Furthermore, based on results of a short-term study performed by our group, that demonstrated an increase in energy expenditure, a positive effect on the regulation of body composition might be expected.

ELIGIBILITY:
Inclusion Criteria:

* Overweight men and women (BMI≥25kg/m2-39.9kg/m2),
* Aged 20-35 and 35-50 years
* Caucasian
* Normal fasting glucose (< 6.1 mmol/L) and normal postprandial glucose (2h-glucose <7.8 mm)
* Normal blood pressure (systolic blood pressure 100-140 mmHg, diastolic blood pressure 60-90 mmHg)
* Weight stable in last 3 months (± 2kg)

Exclusion Criteria:

* Women lactating, pregnant or (post) menopausal
* Regular smokers
* People with intensive fitness training, eg. athletes (≥ 3 per week ≥ 1 hour training)
* Habitual consumption of green tea (more than 1 cup per day) or products containing green tea extract
* Total caffeine consumption > 300 mg/day (1 can of cola or 2 cups of regular coffee or 2 cups of black tea or 1 cup of coffee and 1 cup of black tea or other combinations)
* Alcohol intake >20 g/day (2 glasses of beer or wine)
* Any dietary vitamins or dietary supplements
* Diabetes mellitus (defined as FPG ≥ 7.0 mmol/l and/or 2hPG ≥ 11.1 mmol/l)
* Serious pulmonary, cardiovascular, hepatic or renal disease
* History of cardiovascular disease
* All other relevant medical disorders that potentially interfere with this trial (e.g. history of gastro-intestinal, liver or thyroid disorders)
* Current use of medication interfering with study intervention or interfering with study endpoints/hypotheses (e.g. medication containing caffeine like analgesics, anorectics and analeptics)
* Not to be able to understand the study information
* Subjects on a special diet or vegetarian
* Blood donation 2 months prior to the study and during the study
* Participation in other studies
* Drug use
* Coagulation disorders (i.e. hemophilia (type A, B and C), von Willebrand disease, vitamin K deficiency, afibrinogenemia, disseminated intravascular coagulation and thrombosis)
* Use of anti-coagulant medication
* Acute or history of gastrointestinal diseases (Morbus Crohn, Colitis Ulcerosa)
* Intake of Antibiotics for the last 3 months

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2012-08; Primary Completion 2014-05 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Systemic insulin sensitivity | change from week 0 to week 12 after supplementation
  hyperinsulinemic euglycemic clamp with glucose-tracer

SECONDARY OUTCOMES:
skeletal muscle mitochondrial function | change from week 0 to week 12 after supplementation
  ex vivo skeletal muscle respiratory capacity

OTHER OUTCOMES:
lipid oxidation | change from week 0 to week 12 after supplementation
  fasting and 4-h postprandial (high-fat mixed-meal) by indirect calorimetry
skeletal muscle and adipose tissue lipolysis | change from week 0 to week 12 after supplementation
  microdialysate sample fasting and postprandial (after high-fat mixed-meal)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen E Blaak, Prof., Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University, Maastricht, Netherlands

REFERENCES:
- [Derived] Fazelzadeh P, Hoefsloot HCJ, Hankemeier T, Most J, Kersten S, Blaak EE, Boekschoten M, van Duynhoven J. Global testing of shifts in metabolic phenotype. Metabolomics. 2018 Oct 4;14(10):139. doi: 10.1007/s11306-018-1435-8. PMID 30830386
- [Derived] Most J, Goossens GH, Reijnders D, Canfora EE, Penders J, Blaak EE. Gut microbiota composition strongly correlates to peripheral insulin sensitivity in obese men but not in women. Benef Microbes. 2017 Aug 24;8(4):557-562. doi: 10.3920/BM2016.0189. Epub 2017 Jun 16. PMID 28618864
- [Derived] Most J, Timmers S, Warnke I, Jocken JW, van Boekschoten M, de Groot P, Bendik I, Schrauwen P, Goossens GH, Blaak EE. Combined epigallocatechin-3-gallate and resveratrol supplementation for 12 wk increases mitochondrial capacity and fat oxidation, but not insulin sensitivity, in obese humans: a randomized controlled trial. Am J Clin Nutr. 2016 Jul;104(1):215-27. doi: 10.3945/ajcn.115.122937. Epub 2016 May 18. PMID 27194304